CLINICAL TRIAL: NCT00216879
Title: Long-term Treatment of Scalp Psoriasis With Calcipotriol Plus Betamethasone Dipropionate Gel
Brief Title: Efficacy and Safety of Calcipotriol Plus Betamethasone Dipropionate Gel for up to a Year in Scalp Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MBL 0407 INT
Record Dates: First submitted 2005-09-15; First posted 2005-09-22 (Estimated); Last update posted 2025-02-24 (Actual); Status verified 2015-03

CONDITIONS: Psoriasis of Scalp
MeSH Terms: interventions — calcipotriene

INTERVENTIONS:
Drug: Calcipotriol plus betamethasone dipropionate gel (LEO 80185)

SUMMARY:
The purpose of the trial is to study the safety and efficacy of long term use of once daily applications, as needed, of calcipotriol plus betamethasone dipropionate gel, as compared to calcipotriol alone in the same gel.

The primary response criteria will be the incidence of adverse drug reactions of any type, and the incidence of adverse events of concern associated with long-term corticosteroid use on the scalp.

ELIGIBILITY:
Inclusion Criteria:

* Scalp psoriasis amenable to topical treatment with a maximum of 100 g of study medication per week
* Clinical signs of psoriasis vulgaris on trunk and/or limbs, or earlier diagnosed with psoriasis vulgaris on trunk and/or limbs
* Extent of scalp psoriasis involving more than 10% of the total scalp area
* Disease severity on the scalp graded as Moderate, Severe or Very Severe according to the Investigator's Global Assessment of disease severity

Exclusion Criteria:

* PUVA or Grenz ray therapy anywhere on the patient within 28 days prior to randomisation
* UVB therapy anywhere on the patient within 14 days prior to randomisation
* Systemic use of biological treatments, whether marketed or not, directed against or with a potential effect on, scalp psoriasis (e.g., alefacept, efalizumab, etanercept, infliximab) within 6 months prior to randomisaiton
* Systemic treatments with a potential effect on scalp psoriasis vulgaris (e.g., corticosteroids, retinoids, immunosuppressants) within 28 days prior to randomisation
* Any topical treatment for scalp psoriasis or any other skin disease on the scalp (excluding medicated shampoos, emollients and hair conditioners) within 14 days prior to randomisaiton
* Topical treatment for other skin disorders with very potent WHO group IV corticosteroids within 14 days prior to randomisation
* Planned initiation of, or changes in dose of concomitant medication that could affect scalp psoriasis (e.g., beta blockers, antimalarial drugs, lithium) during the study
* Current diagnosis of guttate, pustular, exfoliative or erythrodermic psoriasis
* Patients with any of the following conditions present on the scalp area: viral lesions, fungal and bacterial skin infections, parasitic infections and atrophic skin
* Known or suspected severe renal insufficiency or severe hepatic disorders
* Patiens with history/signs/symptoms suggestive of an abnormality of calcium homeostasis associated with clinically significant hypercalcaemia
* Trial subjects should be using an adequate method of contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800
Dates: Start 2005-02; Study Completion 2006-07

PRIMARY OUTCOMES:
The proportions of patients who experience adverse drug reactions and the proportion of patients who experience adverse events of concern associated with long-term topical corticosteroid use on the scalp during the study

SECONDARY OUTCOMES:
Percentage of post-baseline satisfactorily controlled assessments according to the Investigators' Global Assessment of disease severity during the study

CONTACTS AND LOCATIONS:
Overall Officials: T A Luger, Dr. med., Principal Investigator — Universitätsklinikum Münster, Klinik und Poliklinik für Hautkrankheiten
Locations (5):
- Clinique de Dermatologie, Moncton, Canada
- Hørsholm Hospital, Dermatological Department, Hørsholm, Denmark
- Hôpital Nord, Service de Dermatologie, Saint-Etienne, France
- Universitätsklinikum Münster, Klinik und Poliklinik für Hautkrankheiten, Münster, Germany
- Monklands Hospital, Department of Dermatology, Airdrie, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Clinical Trials at LEO Pharma — https://www.leopharmatrials.com/en